CLINICAL TRIAL: NCT03567408
Title: Safety and Efficacy of Bivalirudin in Patients With Diabetes Mellitus Undergoing Percutaneous Coronary Intervention (PCI)
Brief Title: Clinical Study of Bivalirudin for Percutaneous Coronary Intervention (PCI)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qian Gong (Other)
Responsible Party: Sponsor-Investigator, Qian Gong, Principal Investigator, Mianyang Central Hospital
Organization: Mianyang Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123456789
Record Dates: First submitted 2018-06-01; First posted 2018-06-25 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective PCI with bivalirudin (Experimental): Before PCI, bivalirudin is intravenously injected with 0.75 mg/kg, 1.75 mg/(kg.h) through continuous intravenous drip to finish surgery (no more than 4 hours), if necessary, after the surgery, with a low dose of 0.2 mg/(kg.h) intravenous drip less than 20 hours.
  Interventions: Procedure: Selective PCI; Drug: Bivalirudin
- Unfractionated heparin (Placebo Comparator): Before PCI, unfractionated heparin sodium is intravenously injected with 70-100 U/kg, and if the operation time exceeded 1h, an additional 1000 U/h would be added.
  Interventions: Procedure: Selective PCI

INTERVENTIONS:
Procedure: Selective PCI — Selective PCI for treatment of elderly patients (age≥65) presenting with diabetes mellitus.
Drug: Bivalirudin — Before, during and after surgery, bivalirudin was used according to the dosage regimen to assess it's impact on elderly patients with diabetes mellitus undergoing selective PCI.
  Other Names: Angiomax
  Arms: Selective PCI with bivalirudin

SUMMARY:
Bivalirudin is widely used as an anticoagulant to reduce the risk of bleeding in PCI perioperative period. Additionally, 15.7%-32.7% patients have diabetes mellitus who undergo percutaneous coronary interventions (PCI), so bivalirudin was used to anticoagulate in these patients to evaluate its safety and efficacy.

DETAILED DESCRIPTION:
Bivalirudin is a specific reversible thrombin direct inhibitor and the function of thrombin activity site can be recovered through hydrolyzing bivalirudin by thrombin. Therefore, bivalirudin is widely used as an anticoagulant during percutaneous coronary intervention (PCI) for coronary heart disease, and 15.7%-32.7% patients have diabetes mellitus who undergo percutaneous coronary interventions (PCI). At the same time, elderly patients have higher risk of bleeding whose age over 65, so bivalirudin can reduce the risk of bleeding and the incidence of net adverse clinical events for the elderly patients whose age over 65 with diabetes mellitus in PCI perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 65 years, with diabetes mellitus.
2. Patients who undergo selective PCI therapy.
3. Patients who agree to participate in this clinical trial and sign informed consent prior to surgery.

Exclusion Criteria:

1. Patients with acute coronary syndrome undergoing primary PCI.
2. Combined with other diseases, the life expectancy of patients don't exceed 1 year.
3. Patients with active bleeding.
4. Bleeding in the gastrointestinal or urogenital tract in the past 6 weeks.
5. Combined with high risk of postoperative hemorrhage, such as active gastric ulcer, active ulcerative colitis, etc.
6. Patients who have undergone major surgery in the last 1 month.
7. A history of intracranial bleeding or structural abnormalities, such as cerebral aneurysms.
8. Patients with cardiogenic shock, or suspected myocarditis, infective endocarditis.
9. Patients who received regular heparin therapy within 6 hours or low molecular weight heparin therapy within 8 hours, or other factors that the researchers believe may influence the outcome of the trial.
10. Patients with severe uncontrolled hypertension.
11. Patients with active hepatitis, HIV and other infectious diseases.
12. Patients with contraindications of bivalirudin and heparin.
13. Other researchers considered the patients are unfit to participate in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2019-08-12 (Estimated); Study Completion 2020-08-12 (Estimated)

PRIMARY OUTCOMES:
activated clotting time(ACT) | 5min after using drug
  The ACT test can be used to monitor anticoagulation effects, such as high-dose heparin before, during, and shortly after procedures that require intense anticoagulant administration, such as cardiac bypass, cardiac angioplasty, thrombolysis, extra-corporeal membrane oxygenation (ECMO) and continuous dialysis

SECONDARY OUTCOMES:
30-day major adverse cardiac events | 30 days
  30-day major adverse cardiac events including recidivation of angina pectoris, in-stent restenosis, severe arrhythmia, cardiac failure, sudden cardiac death.
30-day bleeding events | 30 days
  According to the bleeding academic research consortium (BARC) bleeding classification.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Gong, Master, Study Chair — Mian Yang Central Hospital

IPD SHARING:
Plan to Share IPD: Undecided